CLINICAL TRIAL: NCT07188181
Title: AI and Fluorescence Help Junior Surgeons Identify the Bile Duct During Laparoscopic Cholecystectomy
Brief Title: Using AI and Fluorescence Guidance to Enhance Extrahepatic Bile Duct Identification Among Junior Surgeons During Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202301955B0
Record Dates: First submitted 2025-09-17; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-01

CONDITIONS: Surgical Education and Anatomical Identification in Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; Artificial Intelligence; Common Bile Duct Identification; Indocyanine Green Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PGY Trainees: Postgraduate-year trainees with limited experience in laparoscopic cholecystectomy (<20 cases).
- Junior Residents: Residents with moderate experience in laparoscopic cholecystectomy (20-50 cases)
- Senior Residents: Residents with advanced experience in laparoscopic cholecystectomy (>50 cases).

SUMMARY:
The present study evaluates whether PGY trainees and surgical residents, with or without AI assistance, could accurately identify the presence and anatomical location of the CBD, as well as delineate intraoperative danger zones during LC.

DETAILED DESCRIPTION:
This retrospective cohort study evaluated the impact of artificial intelligence (AI) assistance on anatomical recognition during laparoscopic cholecystectomy (LC). Between June 2022 and December 2024, indocyanine green (ICG) fluorescence-guided LC videos were prospectively collected at a tertiary referral center. After excluding duplicate cases, 177 videos were used for model training, 15 for validation, and 15 for testing. Frames were extracted at 1 frame per second, and key structures including the common bile duct (CBD), cystic duct, cystic artery, liver, gallbladder, and surgical instruments were annotated by board-certified hepatobiliary surgeons to generate the ground truth dataset.

A YOLOv9 object detection model, incorporating Programmable Gradient Information (PGI) and Generalized Efficient Layer Aggregation Network (GELAN), was trained to recognize critical biliary anatomy. For the experimental phase, surgical trainees (postgraduate trainees, junior residents, and senior residents) reviewed condensed 2-3 minute surgical videos, segmented into 5-second clips. In the CBD recognition task, participants determined whether the CBD was visible in each clip. In the CBD annotation task, participants placed bounding boxes to indicate the CBD location on single frames, and additionally delineated a polygonal "dangerous zone" within Calot's triangle where further dissection is considered hazardous.

Each participant first performed both tasks without AI assistance. After a one-week washout, the same tasks were repeated with AI support, which displayed YOLOv9-generated bounding boxes to guide decision-making. The task order was randomized to minimize learning bias. Performance metrics included recognition accuracy, precision, recall, F1-score, and intersection over union (IoU).

This study was retrospectively registered after completion, as it used de-identified surgical videos and trainee assessments.

ELIGIBILITY:
Inclusion Criteria:

* Postgraduate-year (PGY) trainees with fewer than 20 laparoscopic cholecystectomy (LC) cases.
* Junior residents with 20-50 LC cases.
* Senior residents with more than 50 LC cases.

Exclusion Criteria:

* Participants not available for the one-week washout and repeat assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Surgical trainees (postgraduate trainees, junior residents, and senior residents) recruited from a single tertiary academic medical center. Participants performed video-based assessments of indocyanine green-guided laparoscopic cholecystectomy recordings.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
CBD Recognition | During a single video review session (approximately 30-60 minutes per participant)
  identify the presence of the CBD

SECONDARY OUTCOMES:
CBD annotation | During a single video review session (approximately 30-60 minutes per participant)
  Identify the exact location of the CBD

CONTACTS AND LOCATIONS:
Overall Officials: Shih Min Yin, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Shih Min Yin, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because institutional policy prohibits release of de-identified surgical videos and trainee performance data outside the study team.